CLINICAL TRIAL: NCT05773105
Title: Cadonilimab Combined With Regorafenib for Patients With Hepatocellular Carcinoma Who Progressed on Systemic Therapy: An Open Label, Single Arm, Single Center, Prospective, Phase I/II Trial
Brief Title: A Study of Cadonilimab Combined With Regorafenib in Patients With Advanced HCC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhongguo Zhou, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2023-002-01
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: bispecific antibody; advanced HCC; anti-PD-1 and CTLA-4
MeSH Terms: conditions — Diabetes Mellitus, Insulin-Dependent, 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab+regorafenib (Experimental)
  Interventions: Drug: Cadonilimab+regorafenib

INTERVENTIONS:
Drug: Cadonilimab+regorafenib — cadonilimab(10mg/kg, iv,Q3W,D1) + regorafenib(80mg,PO,QD,everyday)

SUMMARY:
To evaluate the efficacy and safety of cadonilimab combined with regorafenib in patients with HCC who progressed on systemic therapy.

DETAILED DESCRIPTION:
Currently, second-line treatment options for advanced HCC (aHCC) patients including single TKI or anti-PD-(L)1 remains limited survival benefits and objective responses. To explore more effective and safer second-line or later therapies for aHCC is necessary. Cadonilimab is a first-in-class humanized IgG1 bispecific antibody that binds to PD-1 and CTLA-4 simultaneously. Dual checkpoint inhibition of the PD-1 and CTAL4 pathways with single cadonilimab has the potential to boost immune surveillance in HCC. Previously data indicated that cadonilimab possesses an encouraging anti-tumour activity and an improved safety profile compared to the co-administration of anti-PD-1 plus anti-CTLA-4 antibodies. Regorafenib is a TKI and approved for second-line treatment of uHCC globally. Here, the investigators evaluated the safety of cadonilimab plus regorafenib as second-line or later therapy in patients with aHCC.

ELIGIBILITY:
Main Inclusion Criteria:

1. Patients who have signed ICF and are able to perform follow-up visits and relevant procedures required in the protocol
2. Age 18-75
3. Histologically or pathologically confirmed hepatocellular carcinoma
4. Barcelona Clinic Liver Cancer (BCLC) stage of B or C or CNLC IIb-IIIb, for those unsuitable for radical surgery and/or local treatment
5. Previously treated with anti-vascular targeting combined with or without anti-PD-1/PD-L1 agents for HCC, with disease progression or intolerable toxicity
6. Child-Pugh score of ≤ 7
7. ECOG PS of 0 or 1
8. At least 1 measurable lesion (according to RECIST1.1)
9. Sufficient organ and bone marrow functions, with the laboratory test values within 7 days before the enrollment meeting the following requirements (no blood components, cell growth factors, albumin, and other drugs via intravenous or subcutaneous administrations are allowed for correction treatment within the first 14 days after the laboratory test results are obtained). The specific information is as follows:

   1. Routine blood test: absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L; platelet count (PLT) ≥ 50× 10^9/L; hemoglobin (HGB) ≥ 9.0 g/dL.
   2. Hepatic function: total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; serum albumin ≥ 28 g/L;
   3. Renal function: serum creatinine (Cr) ≤ 1.5 × ULN or clearance of creatinine (CCr)

      ≥ 60 mL/min (Cockcroft-Gault formula); urinalysis results showing urine protein < 2+; patients whose baseline urinalysis results show urine protein ≥ 2+ should undergo 24-h urine collection and 24-h urine protein quantitation test result should be < 1 g.
   4. Blood coagulation function: international normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
10. Estimated survival ≥ 12 weeks.
11. Female patients of childbearing age or male patients with female sexual partners of childbearing age should take effective contraceptive measures throughout the treatment and 6 months after the last dose

Main Exclusion Criteria:

1. Histologically/cytologically confirmed fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, and cholangiocarcinoma.
2. History of hepatic encephalopathy or liver transplantation.
3. Symptomatic pleural effusion, ascites, and pericardial effusion that require drainage.
4. Acute or chronic active hepatitis B or C infection; hepatitis B virus (HBV) DNA > 2000 IU/mL or 10^4 copies/mL; hepatitis C virus (HCV) RNA > 10^3 copies/mL; hepatitis B surface antigen (HbsAg) and anti-HCV antibody positive concurrently. Those who possess the indicators lower than the above criteria after nucleotide antiviral treatment can be enrolled.
5. Presence of metastasis to the central nervous system.
6. Presence of bleeding events from esophageal or gastric varices caused by portal hypertension within the past 6 months. Presence of known severe (G3) varicose veins in endoscopy within 3 months before the first dose. Evidence of portal hypertension (including the finding of splenomegaly in imaging studies) with a high risk of bleeding assessed by the investigator
7. Presence of any life-threatening bleeding events within the past 3 months, including the need for transfusion, surgery or local treatment, and continuous medication therapy.
8. Any arterial/venous thromboembolic events within 6 months, including myocardial infarction, unstable angina, cerebrovascular accident or transient cerebral ischemic attack, pulmonary embolism, deep vein thrombosis, or any other history of serious thromboembolism. Presence of implantable venous port or catheter-derived thrombosis, or superficial venous thrombosis, barring stable thrombosis following the conventional anticoagulation treatment. Prophylactic use of low-dose low-molecular-weight heparin (e.g., enoxaparin 40 mg/day) is permitted.
9. Involvement of both the main portal vein and the left and right branches by portal vein tumor thrombus, or of both the main trunk and the superior mesenteric vein concurrently. Presence of tumor thrombus of inferior vena cava.
10. Uncontrolled hypertension (systolic greater than 140 mmHg or diastolic greater than 90 mmHg) after the optimal medical treatment, history of hypertensive crisis or hypertensive encephalopathy.
11. Toxicity (excluding alopecia, events not clinically significant, and asymptomatic laboratory abnormalities) caused by previous therapy that has not yet resolved to grade 0 or 1 (National Cancer Institute Common Terminology Criteria for Adverse Events V5.0 (NCI CTCAE V5.0)) before the first dose of study drugs.
12. Symptomatic congestive cardiac failure (NYHA Class II-IV).
13. Serious hemorrhagic tendency or coagulopathy, or currently receiving thrombolytic therapy.
14. History of gastrointestinal perforation and/or fistula, history of bowel obstruction (including incomplete bowel obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection accompanied with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea within the past 6 months.
15. History or current experience of pulmonary fibrosis and such lung diseases as interstitial pneumonia, pneumoconiosis, drug-related pneumonia, and severely impaired lung function.
16. Active or poorly clinically controlled serious infections.
17. Human immunodeficiency virus (HIV) infected (HIV 1/2 antibody positive) and known syphilis infection requiring treatment.
18. Presence of active autoimmune diseases requiring systemic treatment (e.g., use of disease-modifying drugs, corticosteroids, or immunosuppressants) within 2 years before the first dose.
19. Receipt of major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks before the first dose or having unhealed wounds, ulcers, or fractures.
20. Uncontrolled/uncorrectable metabolic disorders, other non-malignant organ diseases, systemic diseases, or cancer-related secondary diseases with the potential to cause a relatively high medical risk and/or survival evaluation uncertainties unsuitable for subject enrollment as judged by the investigator; other circumstances unsuitable for subject enrollment as judged by the investigator.
21. Pregnant or breastfeeding female patients.
22. Acute or chronic diseases, psychiatric disorders, or laboratory abnormalities that may lead to the following consequences: increased study participation or drug-related risks, or interference with interpreting trial results, and considered ineligible for participating in the trial by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Desease control rate (DCR) | At the end of Cycle 2 (each cycle is 21 days)
  Defined as proportion of patients who have CR, PR or SD according to RECIST v1.1

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to two years
  Defined as the time from enrollment to disease progression or death (whichever occurs first)
Overall survival (OS) | Up to two years
  Defined as the time from enrollment to death from any cause
Desease control rate (DCR) | At the end of Cycle 2 (each cycle is 21 days)
  Defined as proportion of patients who have CR, PR or SD according to mRECIST
Adverse Events (AEs) | Up to two years
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No